CLINICAL TRIAL: NCT01318408
Title: A Prospective, Phase 4, Open-Label, Twelve-Week Study to Examine the Cognitive Impact and Tolerability of Levetiracetam (Keppra) in Elderly Patients With Seizures of Partial Onset
Brief Title: Levetiracetam: The Anti-Convulsant of Choice for Elderly Patients With Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEPPRA; WIRB # 20061543 (Other: UCB pharma grant to DUCOM)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levetiracetam (Experimental): Levetiracetam was titrated over 4 weeks, with initial dosing of 250 mg bis in die (BID). Dosing was flexible and was based on the prescribing physician's discretion.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Titration of Keppra will start at 250 mg by mouth twice daily for three days. Then 500 mg by mouth twice daily for three days. Then 750 mg by mouth twice daily for the duration of the study, or for as long as treatment is necessary. This titration schedule is subject to change based on subject's tolerability.
  Other Names: Levetiracetam is the brand name for Keppra

SUMMARY:
Elderly persons with dementia are at risk for seizures, however, traditional anticonvulsants are poorly tolerated in this population. Our goal is to examine Levetiracetam (Keppra) in elderly dementia patients with seizures. While it has been established that Keppra controls seizures in this age group, it is important to demonstrate that treatment with Keppra would not affect cognitive abilities in this large population of patients . As this population is already cognitively impaired, the best choice of anticonvulsant would be one that does not further compromise their cognitive abilities. Keppra is an excellent anticonvulsant agent in the elderly for a variety of reasons, including safety, favorable side effect profile, lack of interaction with other drugs, and efficacy. Our retrospective pilot data suggests that cognition is not negatively affected by Keppra. The current prospective study will assess the cognitive abilities of persons with cognitive impairment at baseline and at weeks 4 and 12. The overall objective is to determine the cognitive tolerability of Keppra for seizures in elderly cognitively impaired patients.

DETAILED DESCRIPTION:
This is a prospective, phase 4, open label, twelve week study. The study will consist of a 4 week titration phase followed by an 8 week assessment phase. All clinic visits will be conducted at Drexel University College of Medicine Department of Neurology at 219 N. Broad St., Phila., PA.

Visit one will include reviewing and signing the written informed consent form, obtaining relevant demographic data, and then routine blood work. The baseline frequency, duration and type of seizures our subjects experience will be documented, as will their current antiepileptic medications. Baseline history and a physical and neurological examination will be performed, including vital signs. Testing will include baseline measurements of cognition, function (activities of daily living), and behavior. Cognitive testing will include Folstein's Minimental State examination (MMSE), and the ADAS-cog. Our overall assessment will include the Modified Schwab and England Activities of Daily Living Scale. Behavioral assessment will include Tariot's Behavior Ratings Scale and the Cohen-Mansfield Agitation Inventory (CMAI; long form). Levetiracetam will be initiated and instructions for follow up will be given. Because the goal is cognitive tolerability, Levetiracetam will be used as either an add-on agent or as primary monotherapy.

During week two, a follow up telephone assessment will be done to review the instructions and to determine whether any medical changes or adverse events occurred. Adverse events will be assessed by direct questioning and spontaneous patient/caregiver reports. The date, number, duration and type of seizures any of our subjects experience will also be documented.

At the third assessment (week 4), a follow up physical and neurological examination will be done, including vital signs, and the mental testing, including the tests of cognition, function and behavior will be repeated. An assessment will be made to determine whether adverse events occurred. Adverse events will be assessed by review of the subject's seizure log, physician observation, direct questioning and spontaneous reports. The date, number, duration and type of seizures any subject experiences will also be documented. In cases where levetiracetam is an add-on agent, we will attempt to taper the preceding medications if seizure control has been demonstrated. Cognitive testing will be done when subjects are not in a post-ictal state. Any subject who has had a seizure with generalization within 24 hours of their scheduled testing will be rescheduled to another day within one week.

At week twelve, a full follow up mental status assessment will be done for the final assessment. Testing will be the same as that done at weeks 1 (baseline) and 4. Again, cognitive testing will not be done when subjects are in a post-ictal state. Any subject who has had a seizure with generalization within 24 hours of their scheduled testing will be rescheduled to the next available day, within one week.

Follow up blood work and a screen for adverse events will also be obtained at that time. Again, adverse events will be assessed by review of their seizure log, physician observation, direct questioning and spontaneous reports. The date, number, duration and type of seizures will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* Meet validated clinical criteria for Alzheimer's disease, mixed dementia or MCI
* Age range greater than or equal to 60 years
* Stable general medical condition as assessed by the investigator
* Seizures which are partial in onset (with or without secondary generalization)
* Subjects with 4 or fewer seizures per month
* MMSE score of less than 28 at baseline
* Patients who are currently being treated with anticonvulsants or those with new onset seizures.

Exclusion Criteria:

* Patients with other clinically significant organic or neurological diseases. Patients considered medically unstable
* Patients in end stage renal disease requiring hemodialysis
* Patients with a known hypersensitivity to Levetiracetam
* Patients with primary generalized epilepsy
* Patients with brain tumors or other significant CNS abnormalities that are the primary cause of the seizures
* Patients with a history of status epilepticus
* Patients with severe psychiatric diagnoses or severe behavioral problems
* Dementia patients lacking a caregiver.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lippa, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine, Dept of Neurology, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Ritchie K, Touchon J. Mild cognitive impairment: conceptual basis and current nosological status. Lancet. 2000 Jan 15;355(9199):225-8. doi: 10.1016/S0140-6736(99)06155-3. No abstract available. PMID 10675135

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: All participants received study drug.
Period: Overall Study
Arm/Group | Open Label
Started | 24
Completed | 16
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 69.9 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: MMSE at Baseline and at Three (3) Months.
Description: The MMSE (Folstein et al 1975) is a brief cognitive test assessing general cognitive function that has been employed in numerous clinical trials of Food and Drug Administration (FDA) products approved for the treatment of AD. The MMSE consists of five components; 1) orientation to time and place, 2) registration of three words, 3) attention and calculation, 4) recall of three words, and 5) language. The scores from each of the five components are summed to obtain the overall MMSE score. The score can range from 0 to 30, with lower scores indicating greater impairment in function.
Time Frame: Baseline and Three months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 24
units on a scale
  Baseline | 18.2 (7.9)
  Change at 3 Months | 2.2 (3.0)
Statistical Analysis 1: Comparison: Open Label; The intent-to-treat group included all individuals who initiated levetiracetam. The Mann-Whitney U test was used to determine changes in participants' scores for cognition, function, and behavior between baseline and 12 weeks.Change in MMSE test scores was the primary outcome measure; Test type: Non-Inferiority or Equivalence — Assessing effects on cognition over time; p = .01, Wilcoxon (Mann-Whitney)

2. Primary Outcome: ADAS-cog at Baseline and at 3 Months.
Description: ADAScog (Alzheimer's Disease Assessment Scale-cognitive subscale) consists of 11 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD. Score ranges from 0 - 70.
  Lower scores (negative change) indicate improvements on the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-cog).
Time Frame: Baseline and Three (3) months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 24
units on a scale
  Baseline | 25.5 (13.8)
  Change at 3 months | -4.3 (6.4)
Statistical Analysis 1: Comparison: Open Label; Test type: Non-Inferiority or Equivalence — Assessing cognitive effects over time; p = .02, Wilcoxon (Mann-Whitney); Lower scores (negative change) indicate improvements on the ADAS-cog

3. Other Pre Specified Outcome: Several Ratings Such as Activities of Daily Living, Behavior and Motor Activity Will Also be Evaluated
Description: Several Ratings Such as Activities of Daily Living, Behavior and Motor Activity Were Planned to be Examined.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: study was conducted for 12 weeks with an 8 week follow up
Groups:
- Open Label: All participants received study drug. Four withdrew due to adverse events; related to fatigue.
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (N=24)
fatigue (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No